CLINICAL TRIAL: NCT02539069
Title: A Post-marketing Surveillance to Evaluate the Efficacy and Safety of CHONDRON (Autologous Cultured Chondrocyte) Through Arthroscopy in Patients With Knee Cartilage Defects
Brief Title: The Post-marketing Surveillance to Evaluate the Efficacy of CHONDRON (Autologous Cultured Chondrocyte) by Arthroscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sewon Cellontech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09CON
Record Dates: First submitted 2015-08-28; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Osteoarthritis; Traumatic Arthritis
Keywords: cartilage defects; Chondron; Autologous cultured Chondrocyte; arthroscopy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chondron Implantation (Experimental): Chondron Implantation for the suject with cartilage defect through arthroscopy
  Interventions: Device: Chondron Implantation

INTERVENTIONS:
Device: Chondron Implantation — In one vial (0.4 ml), Main ingredient: 1.2 million or more autologous chondrocytes Culture solution: Adequate amount of Dulbecco's modified Eagle medium (DMEM) The cells that fill the vial are sufficiently suspended, and a sufficient amount of suspension is grafted in the defect with fibrin glue.

SUMMARY:
A clinical trial to evaluate the long-term efficacy and safety of Chondron (Autologous cultured Chondrocyte) administered through arthroscopy from the drug's 48 weeks efficacy and safety evaluation with 96 weeks follow-up in patients with knee cartilage defects.

DETAILED DESCRIPTION:
This is an open trial, involving a total of 10 subjects. Subjects who give consent will be screened and those who meet trial criteria will receive CHONDRON (Autologous cultured Chondrocyte) by transplant. During the trial period, subjects must follow the instructions given by principal investigator. Subjects will make 8* hospital visits on a regular basis inclusive of hospitalization. During these visits subjects will be examined. For the evaluation of safety and efficacy of CHONDRON, examination with doctors, blood samples, x-ray, MRI tests, observation with the naked eyes and arthroscopy will be performed. *If tissue samples can be collected at screening visit, there will be only 7 visits.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cartilage defects in their knee (Including Knee OA and Knee TA) * For a single lesion, less than 15 cm2 cartilage defects; and for multiple lesions, less than 20 cm2
2. Patients with misalignment of their tibia and femur, unstable ligament in their knee, or bony defects in the lesions of their knee, and/or who had been treated for alignment
3. Patients which surrounding cartilage are normal
4. Patients who were 15 years old or older
5. Patients or their representative (for adults), or patients and their parent/guardian (for minors), who agreed to participate in the study and signed the informed consent form

Exclusion Criteria:

1. Patients hypersensitive to bovine protein
2. Patients hypersensitive to gentamicin antibiotics
3. Patients with inflammatory arthritis such as rheumatoid arthritis, gout arthritis
4. Patients with arthritis related to autoimmune disease
5. Pregnant, breast-feeding patients or those who have a possibility of pregnancy
6. Patients with accompanying diseases other than articular cartilage defects, including tumors (Exception: if the possibility of Chondron treatment is confirmed with doctor's clinical decision).
7. Patients who have a history of receiving radiotherapy, chemotherapy in the last 2 years (Exception: if the possibility of Chondron treatment is confirmed with doctor's clinical decision).
8. Patients with diabetes (however, patients whose blood sugar test results are normal and do not have any complication of diabetes, when a written opinion that CHONDRON administration is possible is appended by a doctor are excluded)
9. Patients with an infection that required hospitalization for antibiotics or the administration of antiseptic agents
10. Patients under adrenocorticoid therapy (Exception: if the possibility of Chondron treatment is confirmed with doctor's clinical decision).
11. Patients with psychiatric disorder and those who are considered to be inappropriate for this trial by the judgment of the clinical trial manager
12. Patients with cartilage defects in both knees (If the necessity of other surgery on the opposite side of knee joint using Chondron is confirmed with doctor's clinical decision).
13. Patients with liver, heart, or kidney disease (Those who show normal or insignificant test results may be enrolled in this study and receive the Chondron based on the investigator's judgment. Hypertension patients are allowed.)
14. Patients who had been infected with a virus (Those who show normal or insignificant test results may be enrolled in this study and receive the Chondron based on the investigator's judgment.)
15. Patients who had participated in another clinical trial (limited to those who participated in other studies on fracture within the last six months.)

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-02 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
change in pain of 100mm Visual Analog Scale | 48 weeks after the surgery
  The primary endpoint for the analysis is the change in the 100mmVAS at 48 weeks after the surgery compared to that at baseline.

SECONDARY OUTCOMES:
change of IKDC (International Knee Documentation Committee) | baseline and 48 weeks after the surgery and 12, 24 and 96 weeks after the surgery
  The IKDC values of the affected knee at baseline and 48weeks after the surgery will be primarily compared based on the evaluations by the subjects and the investigators (and 12, 24 and 96 weeks after the surgery).
Chnage of KSS(Knee Society Score) | baseline and 48 weeks after the surgery and 12, 24 and 96 weeks after the surgery
  The primary endpoint for the analysis is the change in the KSS before and 48 weeks after the surgery (and 12, 24 and 96 weeks after the surgery).
Chnage of ICRS(International Cartilage Repair Society) score | baseline and 48 weeks after the surgery
  The ICRS grades of the affected knee at baseline and 48 weeks after the surgery will be primarily compared.
Chnage of KOOS(Knee injury and osteoarthritis outcome) score | baseline and 48weeks after the surgery and 12, 24 and 96 weeks after the surgery
  The primary endpoint for the analysis is the change in the KOOS at baseline and 48 weeks after the surgery (and 12, 24 and 96 weeks after the surgery).
Change of MRI and mMOCART result | baseline and 48 weeks after the surgery and 12, 24 and 96 weeks after the surgery
  The morphological improvement from MRI iamge of affected knee will be assessed at 48 weeks after the surgery from image at baseline (and 12, 24, and 96 weeks after the surgery). The primary endpoint for the analysis is the change in the mMOCART at baseline and 48 weeks after the surgery (and 12, 24 and 96 weeks after the surgery).
change in pain of 100mm Visual Analog Scale | baseline and 12, 24 and 96 weeks after the surgery
  The change in the 100mmVAS at baseline, 12, 24 and 96 weeks after the surgery will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Jae Kim, MD, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Severance Hospital, Seoul, Seoul, South Korea